CLINICAL TRIAL: NCT05684744
Title: Roflumilast Versus Methotrexate in the Treatment of Psoriasis
Brief Title: Roflumilast Versus Methotrexate in Psoriasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Saadi, Associate Professor of Dermatology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kapu27
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Roflumilast; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Roflumilast (Experimental): oral roflumilast in a dose of 500 mcg per day
  Interventions: Drug: Roflumilast
- Methotrexate (Active Comparator): oral methotrexate in a dose of 0.2- 0.4 mg/kg/week
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Roflumilast — The patients will receive oral roflumilast in a dose of 500 mcg per day for 12 weeks
  Other Names: Roflumilast oral
  Arms: Roflumilast
Drug: Methotrexate — The patients will receive methotrexate in a dose of 0.2- 0.4 mg/kg/week for 12 weeks
  Other Names: Methotrexate tablets
  Arms: Methotrexate

SUMMARY:
Roflumilast is a phosphodiesterase-4 (PDE-4) inhibitor, which is approved in its oral form for chronic obstructive pulmonary disease, and in its topical form in the treatment of plaque psoriasis. Methotrexate is one of the conventional systemic treatments of psoriasis, so the aim of this study is to compare the efficacy and safety of roflumilast and methotrexate in the treatment of psoriasis

DETAILED DESCRIPTION:
Phosphodiesterase (PDE-4) activity was found to be greater in psoriatic skin than in healthy skin. Inhibition of PDE-4 inhibits the hydrolysis of cyclic AMP in inflammatory cells, which increases intracellular cAMP and results in down-regulation of immune modulators, including tumor necrosis factor (TNF)- α, interferon-γ, interleukin (IL)-17, and IL-23. Roflumilast is a potent and selective inhibitor of PDE-4 which is already approved in its oral form for chronic obstructive pulmonary disease. Regarding Roflumilast's topical form, it is currently also approved in the treatment of psoriasis. Lebwohl et al., 2020 found that roflumilast cream was efficacious in reducing the severity of psoriasis in a 12-week, randomized, double-blind, placebo vehicle-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with psoriasis vulgaris
2. Psoriatic patients not receiving any relevant systemic treatment for at least 4 weeks before initiation of our study
3. Psoriatic patients not receiving any relevant topical treatment for at least 2 weeks before initiation of our study

Exclusion Criteria:

1. Erythrodermic or pustular psoriasis
2. Pregnant and lactating females
3. Patients with autoimmune diseases e.g. systemic lupus erythematosus
4. Patients with solid or hematological malignancies e.g., breast cancer, leukemia, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-14 (Actual)

PRIMARY OUTCOMES:
Psoriasis Severity Index (PASI) before and after Roflumilast | 12 weeks
  Comparison of Psoriasis Severity Index (PASI) before and after treatment with Roflumilast, where the lower score indicates clinical improvement. PASI score ranges from 0-72.
Psoriasis Severity Index (PASI) change with Roflumilast Vs Methotrexate | 12 weeks
  Comparison of change of Psoriasis Severity Index (PASI) after treatment with roflumilast and after treatment of methotrexate where the lower score indicates clinical improvement. PASI score ranges from 0-72.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No